CLINICAL TRIAL: NCT01686672
Title: Web-based Delivery of Effective Treatment for Growth in Cystic Fibrosis
Acronym: Be In Charge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-0467
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Behavioral Intervention; Children
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fees and Charges

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web Intervention (Experimental): BeInCharge has two components: an electronic diet tracker and a 7 session intervention. The 7 treatment sessions are designed to be completed over a 7 to 10 week period. Each treatment module includes both a nutrition education and child behavior management component. Treatment sessions should be completed every 7 to 10 days, while the electronic diet tracker requires daily input.
  Interventions: Behavioral: Web Intervention
- Usual Care (No Intervention): Participants will receive usual care and be assessed at baseline and week 10 for study outcomes.

INTERVENTIONS:
Behavioral: Web Intervention — Behavioral
  Other Names: Be In Charge
  Arms: Web Intervention

SUMMARY:
This study will demonstrate feasibility and collect pilot data via a pilot randomized trial of 20 participants on the effectiveness of a web-based delivery system of behavioral plus nutrition intervention for parents of children with Cystic Fibrosis (CF) ages 4 to 9 years of age that has been found to be efficacious in face to face delivery.

DETAILED DESCRIPTION:
Optimizing nutritional status and growth improves health outcomes and survival in children with cystic fibrosis (CF). Better pulmonary function, as measured by forced expiratory rate in 1 second (FEV1), is associated with body mass index (BMI) above the 50th percentile for age and gender for children with CF1. Evidence based practice guidelines recommend that nutritional treatment for children with CF ages 2 to 20 years should aim to achieve and maintain a BMI > 50th percentile, however across 117 CF centers in the United States 57% of girls and 56% of boys failed to meet this recommendation1. The investigators have developed a highly effective behavioral plus nutrition intervention (BE IN CHARGE) and demonstrated its efficacy when delivered face-to-face to produce weight gain and its superiority over nutrition education alone. Although endorsed by the CF Foundation as an evidence-based treatment, it is not available to most CF Centers or families due to lack of trained personnel, cost, and distance issues. With funding from the CF Foundation the investigators developed a web-based delivery system of their efficacious behavioral plus nutrition intervention for parents of children with CF ages 4 to 9 years of age. Using a Place Outcomes Award the investigators have conducted beta testing of the web-intervention and made appropriate modifications. The current study represents the next steps in refining and testing our web-based intervention. This study will demonstrate feasibility and collect pilot data on the effectiveness of the intervention in a pilot randomized trial of 20 treatment naïve participants.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cystic Fibrosis
* Ages 4 to 9 year
* below the 50th percentile for body mass index for age and gender
* and their parents

Exclusion Criteria:

* medical condition that would affect diet or growth (e.g., type 1 diabetes mellitus)
* significant developmental delays
* a sputum culture positive for Burkholderia cepacia
* a forced expiratory volume in the first second of expiration (FEV1) of less than 40%
* receiving enteral or parenteral nutrition.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Average Daily Caloric Intake | Baseline and 10 weeks
  Change in average daily caloric intake at baseline and 10 weeks.

SECONDARY OUTCOMES:
Change in Weight | Baseline and 10 weeks
  Change in weight from baseline to 10 weeks

OTHER OUTCOMES:
Use of web-based intervention | 10 weeks
  Ongoing use of web-intervention collected electronically via the web to include sign on, duration of time on web, page views, and completion of activities on the web-site
Treatment Satisfaction | 10 weeks
  Assessment of participant's satisfaction with the intervention and web-site

CONTACTS AND LOCATIONS:
Overall Officials: Lori Stark, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States